CLINICAL TRIAL: NCT02585336
Title: Effects of Sugar-sweetened Beverage Consumption Changes on Metabolic Health: Improving Metabolic Profile Very Effortlessly (IMPROVE)
Brief Title: Changes in Sugar-sweetened Beverage Intake and Metabolic Health: Improving Metabolic Profile Very Effortlessly
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-16880
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Metabolic Health
Keywords: Sugar-Sweetened beverages; Metabolic health; Soft drinks
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention)
- Brief intervention (Experimental)
  Interventions: Behavioral: Brief intervention

INTERVENTIONS:
Behavioral: Brief intervention — An interviewer provides health information, elicits motivation to reduce SSB consumption, and helps participants make implementation plans. Booster phone calls occur at 1 week after the intervention visit, and at 2 weeks and 24 weeks following the date on which SSBs sales ended at the participant's work location.
  Arms: Brief intervention

SUMMARY:
Sugar-sweetened beverages (SSBs) have been epidemiologically linked to serious health problems including heart disease, liver disease, and diabetes. This study will recruit frequent SSB drinkers who are employees at the University of California, San Francisco (UCSF) and measure markers of metabolic health on two occasions, 10 months apart. During this time, UCSF will cease selling SSBs at all campus and medical center locations. Additionally, at the first assessment half of participants will be randomly assigned to a brief intervention to help reduce SSB consumption, consisting of a 10-20 minute semi-structured interview designed to share health information about SSBs, elicit motivations to reduce consumption, and help set concrete plans to reduce consumption. The investigators will be able to compare changes in metabolic health among those who do and do not reduce SSB consumption. This will make a unique contribution to the growing evidence regarding both the effects of SSB consumption on health and the modifiability of SSB-related health conditions.

DETAILED DESCRIPTION:
Sugar-sweetened beverages (SSBs) have been epidemiologically linked to serious health problems including heart disease, liver disease, and diabetes. This study will recruit frequent SSB drinkers who are employees at the University of California, San Francisco (UCSF) and measure markers of metabolic health on two occasions, 10 months apart. During this time, UCSF will cease selling SSBs at all campus and medical center locations. Additionally, at the first assessment half of participants will be randomly assigned to a brief intervention to help reduce SSB consumption, consisting of a 10-20 minute semi-structured interview designed to share health information about SSBs, elicit motivations to reduce consumption, and help set concrete plans to reduce consumption. We will be able to compare changes in metabolic health among those who do and do not reduce SSB consumption. This will make a unique contribution to the growing evidence regarding both the effects of SSB consumption on health and the modifiability of SSB-related health conditions.

Two key clarifications about the design of this study:

1. The cessation of sugar-sweetened beverage sales is a pre-existing workplace initiative. This study is taking advantage of its initiation but it is not part of the study intervention.
2. The primary predictor in this study is SSB consumption, not condition assignment. Although we will report on the efficacy of the brief intervention, the main goal of the study is to examine the correlational relationship between changes in SSB consumption and changes in health, whether the reduction is associated with the intervention or with other factors.

Planned analyses:

1. For all outcomes other than sugar consumption and SSB consumption (see below), the primary analytic strategy will be to correlate changes in SSB consumption with changes in the outcome.
2. We will additionally assess the efficacy of the university initiative and the brief counseling intervention using a linear mixed regression model estimating the effects of 1) time (pre to post), representing the effect of the university SSB initiative, and 2) assignment to the brief intervention interacting with time.

For both types of analysis, we will include demographic and job-related covariates based on fit criteria to guide model selection.

ELIGIBILITY:
Inclusion Criteria:

* Employed at UCSF
* Reports drinking an average of 60oz or more of sugar-sweetened beverages per week (approximately 8oz/day), over the past month.

Exclusion Criteria:

* Unwilling or medically advised not to fast in preparation for a fasting blood draw
* Reports vasovagal response (fainting) following blood draws or needle sticks in the past.
* Pregnant (health outcome measures from pre- to post-partum will not be comparable).
* Diagnosed with diabetes (type 1 or type 2)
* Not fluent in English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2016-10-16 (Actual); Study Completion 2016-10-16 (Actual)

PRIMARY OUTCOMES:
Homeostatic Model Assessment ratio (HOMA) | 10 month minus baseline
  insulin sensitivity measure derived from fasting glucose and insulin

SECONDARY OUTCOMES:
Waist-hip circumference ratio | 10 month minus baseline
  A measure of abdominal adiposity
Consumption of sugar-sweetened beverages | 2 weeks post-SSB sales ban (1-3 months after initial visit) minus baseline
  outcome for intervention efficacy analysis only

OTHER OUTCOMES:
Reward-based eating drive | 10 month minus baseline
  self-report measure of hedonic drive in eating
Consumption of sugar-sweetened beverages | 10 month minus baseline
  In most analyses treated as a predictor, but used as an outcome when testing the efficacy of the intervention
Total dietary sugar consumption | 10 month minus baseline
  In most analyses treated as a predictor, but used as an outcome when testing the efficacy of the intervention
Glycated hemoglobin (HbA1c) | 10 month minus baseline
  Indicator of long-term glycemic control
Fasting triglycerides | 10 month minus baseline
  Marker of metabolic health and cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Epel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Share database on open science framework.
Supporting Information: Study Protocol, ICF
Time Frame: 5 years
Access Criteria: Deidentified participant data open to all researchers.
URL: https://osf.io/

REFERENCES:
- [Result] Epel ES, Hartman A, Jacobs LM, Leung C, Cohn MA, Jensen L, Ishkanian L, Wojcicki J, Mason AE, Lustig RH, Stanhope KL, Schmidt LA. Association of a Workplace Sales Ban on Sugar-Sweetened Beverages With Employee Consumption of Sugar-Sweetened Beverages and Health. JAMA Intern Med. 2020 Jan 1;180(1):9-16. doi: 10.1001/jamainternmed.2019.4434. PMID 31657840
- [Derived] Wojcicki JM, Lustig RH, Jacobs LM, Mason AE, Hartman A, Leung C, Stanhope K, Lin J, Schmidt LA, Epel ES. Longer Leukocyte Telomere Length Predicts Stronger Response to a Workplace Sugar-Sweetened Beverage Sales Ban: An Exploratory Study. Curr Dev Nutr. 2021 May 26;5(7):nzab084. doi: 10.1093/cdn/nzab084. eCollection 2021 Jul. PMID 34235373
- [Derived] Mason AE, Schmidt L, Ishkanian L, Jacobs LM, Leung C, Jensen L, Cohn MA, Schleicher S, Hartman AR, Wojcicki JM, Lustig RH, Epel ES. A Brief Motivational Intervention Differentially Reduces Sugar-sweetened Beverage (SSB) Consumption. Ann Behav Med. 2021 Oct 27;55(11):1116-1129. doi: 10.1093/abm/kaaa123. PMID 33778854